CLINICAL TRIAL: NCT03265899
Title: Double-blind, Placebo-controlled, Randomized Study: Oxytocin Modulation of Stress-Associated Chemosignals Processing
Brief Title: Oxytocin and the Processing of Social Stress-Associated Chemosignals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Prof. Dr. Dr., University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OXT_OLF_2017
Record Dates: First submitted 2017-08-18; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): 40 IU Oxytocin, intranasal application 30 min prior to the experiment
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): sodium chloride solution, intranasal application 30 min prior to the experiment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40 IU; 5 puffs balanced across nostrils, at an inter-puff interval of 30 seconds
  Other Names: Syntocinon-Spray, Novartis
  Arms: Oxytocin
Drug: Placebo — Placebo nasal spray, 5 puffs balanced across nostrils, at an inter-puff interval of 30 seconds
  Other Names: Placebo-Spray, Novartis
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oxytocin modulates the processing of stress-associated chemosignals and which substrates are involved.

DETAILED DESCRIPTION:
Social transmission of stress and fear is not restricted to visual or auditory cues, but extends to the olfactory domain, a phylogenetically more ancient sense. Exposure to axillary sweat from healthy volunteers undergoing an emotional stressor task evokes a strong vicarious stress response on the behavioral and neural level.Particularly, anxious individuals have been shown to exhibit a heightened sensitivity to social chemosensory stress cues (axillary sweat). The neuropeptide oxytocin (OXT) exerts anxiolytic and anti-stress effects in visual and auditory modalities, however, it still elusive whether OXT also modulates the processing of stress-associated chemosignals. Axillary sweat were obtained from an unrelated sample of 30 healthy men undergoing the Trier Social Stress Test and ergometer training as control.Subsequently, subjects completed a forced-choice emotional face recognition task composed of stimuli with varying intensities (neutral to fearful), while they were exposed to both sweat stimuli and a non-social control odor (raspberry) after OXT or placebo administration, respectively. The investigators expect that OXT selectively diminishes chemosensory-induced behavioral biases and neural responses to stress-related odors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Right-handed

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Tobacco smokers
* MRI contraindications (e.g. metal in body, claustrophobia)
* Anosmia
* Medication known to interfere with olfactory processing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Forced-choice ratings of morphed emotional faces with varying intensities (neutral to fearful). | 30 min after nasal spray administration
  After each trial, subjects were asked to use a button response grip to indicate whether they perceived the depicted face as neutral or fearful.
Response time for facial stimuli ratings. | 30 min after nasal spray administration
Blood-oxygen-level dependent signal in response to chemosensory cues. | 30 minutes after nasal spray administration
  The modulatory effect of oxytocin on neural correlates Using functional magnetic resonance imaging, signal changes in the amygdala, hippocampus and the anterior cingulate cortex in response to olfactory cues of stress and sport (axillary sweat obtained from an unrelated sample of 30 healthy men undergoing the Trier Social Stress Test and ergometer training as control).

SECONDARY OUTCOMES:
Questionnaire measurement of mood (PANAS). | 15 minutes before the nasal spray administration and (on average) 10 minutes after the fMRI experiment
Saliva oxytocin concentrations | immediately before the nasal spray administration and (on average) 10 minutes after the fMRI experiment
Questionnaire measurement of anxiety (STAI). | 15 minutes after nasal spray administration and (on average) 10 minutes after the fMRI experiment

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc MD PhD, Principal Investigator — Department of Psychiatry, University of Bonn, Germany

IPD SHARING:
Plan to Share IPD: No